CLINICAL TRIAL: NCT06316622
Title: Examination of the Relationship Between Body Mass Index and the Skin-epidural Space Distance Measured by Ultrasound in the Lumbar Region
Brief Title: Examination of The Relationshıp Between Body Mass Index And The Skin-Epidural Space Distance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Kaytancı, Principal Investigator, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/08/42
Record Dates: First submitted 2024-02-19; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia Awareness
MeSH Terms: conditions — Intraoperative Awareness | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: relationship between body mass index and the skin epidural space distance
Masking Description: relationship between body mass index and the skin epidural space distance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteer person (Experimental): meausered by ultrasound
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — measured by ultrasound

SUMMARY:
Aim: The aim of the study; to investigate whether there is a relationship between body mass index (BMI), waist circumference, and abdominal subcutaneous adipose tissue and the skin-epidural space distance measured by USG.

DETAILED DESCRIPTION:
The research was carried out in the block room in the preoperating room of Dokuz Eylül University Practice and Research Hospital and with 42 volunteer operating room workers aged between 18-59 years. Height, weight and waist circumference measurements were made with standard measuring instruments, and other measurements were completed by ultrasonography (USG) separately by an anesthesiologist and a radiologist. For ultrasonographic evaluation, left lateral decubitus, right lateral decubitus and in sitting position, skin-dural junction, skin-vertebra corpus, anterior complex distances, upper and lower SIAS levels were examined with convex probe as transverse median. In addition, abdominal subcutaneous fat thickness measurements were made with a linear probe in the supine position. The statistical correlations of all measurements were examined.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 59 years old.
2. ASA I-II classification.
3. Body Mass Index (BMI): 18.5-29.9 kg/m2.

Exclusion Criteria:

1. Individuals under 18 or over 59 years old.
2. Those with a history of vertebral surgery.
3. Patients diagnosed with spinal deformities (excluding scoliosis ≤10 degrees, kyphosis <30 or >80 degrees).
4. Individuals with rheumatologic diseases affecting skeletal structure such as ankylosing spondylitis, rheumatoid arthritis.
5. Presence of wounds or infections in the lumbar region.
6. Volunteers who underwent epidural or spinal interventions in the lumbar region within the last month.
7. Individuals with bone implants affecting posture, such as hip or knee prostheses.
8. Pregnant women.
9. Individuals with conditions like Cushing's syndrome, hypothyroidism, acromegaly causing lumbar edema.
10. Volunteers using corticosteroids.
11. Obese individuals (BMI: >29.9).

Ages: 21 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
We examined the relationships between body mass index calculated by measuring weight and height, subcutaneous fat tissue in the abdominal region and the skin-epidural space distance in the lumbar region; measured by ultrasound. | six months
  Unexpectedly low skin-epidural space distances can be seen even in individuals with high weight and fat content.
  For the targeted space between above the anterior superior iliac spine (ASIS) (estimated L3-L4) and below the ASIS, each patient was positioned in the left lateral, right lateral and then sitting positions, with a transverse-median approach performed by an anaesthetist followed by a radiologist. Skin-dural composite (SDC), skin-vertebral body and anterior complex (posterior longitudinal ligament) distance measurements were recorded separately. Subcutaneous abdominal fat thickness was measured using a linear probe of an ultrasound device (LOGIQ-E, GE Medical Systems, China) to ensure consistency. Measurements were taken at two points (right lateral, left lateral) 2 cm away from the umbilicus and recorded by averaging. Waist circumference was measured using a standard measuring tape at the navel level in all volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Küçükgüçlü, doctor, Study Chair — Dokuz Eylul University
Locations (2):
- Turkey (Türkiye) (2):
  - Dokuz Eylul Unicersity, Izmir, Narlidere
  - Dokuz Eylul University, Izmir